CLINICAL TRIAL: NCT06580821
Title: Evaluation of the Efficacy of the Modified Free Gingival Graft Technique
Brief Title: Efficacy of the Modified Free Gingival Graft Technique
Acronym: FGG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Especialidades Espiritu Santo (Other)
Responsible Party: Principal Investigator, Antonio Lanata Flores, Assistant Professor, Universidad de Especialidades Espiritu Santo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-ODONT-002A
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Modified Free Gingival Graft , Connective Tissue Graft
Keywords: Gingival Recession; Surgical Flaps; Connective Tissue
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial will performed in 30 patient with RT1 gingival recessions at mandibular incisors
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will not know which technique is being used to treat gingival recession.
  The investigator will not be informed which cover up treatment was performed in the gingival recession.
  The outcomes assessor will not be informed of which procedures were performed on the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified free gingival graft (Experimental)
  Interventions: Procedure: mucogingigval surgery
- Conventional free gingival graft (Active Comparator)
  Interventions: Procedure: mucogingigval surgery

INTERVENTIONS:
Procedure: mucogingigval surgery — Is a form of mucogingival surgery that attempts to improve the height of the keratinized tissue (KT), as well as augment the thickness of the gingival phenotype to facilitate meticulous oral hygiene.

SUMMARY:
Gingival recessions can be defined as the exposure of the root surface after an apical migration of the gingival margin in relation to the cemento-enamel junction. Gingival recessions affect both younger and older populations. Various surveys revealed that 88% of people ≥65 years of age and 50% of people between 18 and 64 years of age have ≥1 site with gingival recession. Gingival recessions can occur due to anatomical, pathological factors or trauma and will result in a loss of attachment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least two or less localized recession in mandibular incisors
* Cairo type 1 recession
* Patients who have good plaque control of less than 20%
* Patients between 18-64 years old

Exclusion Criteria:

* Systemically compromised patients
* Smoker patients
* Pregnant women, breastfeeding or use of oral contraceptives
* Patients who are taking medication that may affect healing and coagulation
* Previous periodontal surgeries in the RG area
* Patients with periodontal disease
* Patients who have undergone chemotherapy and radiotherapy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term efficacy of the modified free gingival graft technique on root coverage. | From enrollment to the end of treatment at 12 months, evaluating at 7 days, 14 days, at the first month and after that every 3 months.
  This technique is a modified version of the Free gingival graft, which is a surgery that attempts to improve the height of the keratinized tissue, as well as augment the thickness of the gingival phenotype. This modified version is based on a connective pedicle flap is flipped from its apical origin to cover the exposed root surface prior to the positioning of the Free gingival Graft. The rationale behind the approach is to improve the revascularization of the graft.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidadees, Samborondón, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carcuac O, Trullenque-Eriksson A, Derks J. Modified free gingival graft technique for treatment of gingival recession defects at mandibular incisors: A randomized clinical trial. J Periodontol. 2023 Jun;94(6):722-730. doi: 10.1002/JPER.22-0581. Epub 2023 Jan 30. PMID 36627509